CLINICAL TRIAL: NCT03778775
Title: Transient Elastography (FibroTouch) for Assessing Risk of Gastroesophageal Varices Bleeding in Patients With Compensated Cirrhosis (Pan-CHESS1801): An International Multicenter Study
Brief Title: Transient Elastography (FibroTouch) for Assessing Risk of Gastroesophageal Varices Bleeding in Compensated Cirrhosis (Pan-CHESS1801)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Beijing Tsinghua Changgeng Hospital (Other); LanZhou University (Other); Beijing 302 Hospital (Other); Xijing Hospital of Digestive Diseases (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Zhujiang Hospital (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); The Central Hospital of Lishui City (Other); Xingtai People's Hospital (Other); Seventh Medical Center of PLA Army General Hospital (Other); Shandong Provincial Hospital (Other Government); Southern Medical University, China (Other); Medistra Hospital, University of Indonesia (Unknown); Ankara University (Other); Osaka City University (Other); Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Director, Hepatic Hemodynamic Lab, Nanfang Hospital, Southern Medical University
Other Study IDs: Pan-CHESS1801
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Compensated Liver Cirrhosis; Gastroesophageal Varices Bleeding
Keywords: Transient elastography; Gastroesophageal varices bleeding; Varices needing treatment
MeSH Terms: interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overall eligible participants: Eligible participants will receive standard esophagogastroduodenoscopy and liver stiffness measurement by FibroTouch.
  Interventions: Diagnostic Test: Liver sitffness measurement

INTERVENTIONS:
Diagnostic Test: Liver sitffness measurement — Liver sitffness measurement is performed by FibroTouch, a new-generation of transient elastography with the tesing interval between liver sitffness measurement and esophagogastroduodenoscopy less than one week.
  Other Names: Esophagogastroduodenoscopy

SUMMARY:
Gastroesophageal varices occurs in approximately half of the patients with liver cirrhosis. Variceal bleeding is the most common lethal complication directly from cirrhotic portal hypertension. The golden standard for diagnosing gastroesophageal varices and evaluating the risk of variceal bleeding is the esophagogastroduodenoscopy. According to the Baveno VI consensus, for those with high-risk varices (varies needing treatment), either non-selective beta blockers or endoscopic band ligation is recommended for the prevention of the first variceal bleeding. However, the invasiveness and uncomfortableness during the esophagogastroduodenoscopy procedure has hindered its routine use in clinical practice, especially in compensated cirrhotic patients.

The important role of transient elastography for defining the presence of high-risk varices was highlighted in the Baveno VI consensus workshop that cirrhotic patients with a liver stiffness measurement (LSM) of less than 20 kPa and a platelet count of greater than 150,000/μL can avoid screening endoscopy. In addition, transient elastography-based models (e.g. LSM combined with platelet count, liver stiffness spleen diameter-to-platelet score) were shown to have potentials in distinguish the absence of high-risk gastroesophageal varices. However, this cutoff value of LSM was validated mainly in cohorts with alcoholic or hepatitis C virus dominated cirrhosis. The unmet need is a precise cutoff to rule out high-risk varices in hepatitis B virus dominated cirrhosis, which is an outstanding issue in Asia-Pacific population.

FibroTouch (Hisky Medical Technologies Co. Ltd, Wuxi, China) is a new-generation of transient elastography based on a two-dimensional image-guided system to ensure the precise orientation. In the present study, the investigators aim to conduct an international prospective diagnostic trial with 16 sites to develop and validate the diagnostic performance of FibroTouch-based models for assessing risk of gastroesophageal varices bleeding in compensated cirrhosis.

DETAILED DESCRIPTION:
Gastroesophageal varices occurs in approximately half of the patients with liver cirrhosis. Variceal bleeding is the most common lethal complication directly from cirrhotic portal hypertension. The golden standard for diagnosing gastroesophageal varices and evaluating the risk of variceal bleeding is the esophagogastroduodenoscopy. According to the Baveno VI consensus, for those with high-risk varices (varies needing treatment), either non-selective beta blockers or endoscopic band ligation is recommended for the prevention of the first variceal bleeding. However, the invasiveness and uncomfortableness during the esophagogastroduodenoscopy procedure has hindered its routine use in clinical practice, especially in compensated cirrhotic patients.

The important role of transient elastography for defining the presence of high-risk varices was highlighted in the Baveno VI consensus workshop that cirrhotic patients with a liver stiffness measurement (LSM) of less than 20 kPa and a platelet count of greater than 150,000/μL can avoid screening endoscopy. In addition, transient elastography-based models (e.g. LSM combined with platelet count, liver stiffness spleen diameter-to-platelet score) were shown to have potentials in distinguish the absence of high-risk gastroesophageal varices. However, this cutoff value of LSM was validated mainly in cohorts with alcoholic or hepatitis C virus dominated cirrhosis. The unmet need is a precise cutoff to rule out high-risk varices in hepatitis B virus dominated cirrhosis, which is an outstanding issue in Asia-Pacific population.

FibroTouch (Hisky Medical Technologies Co. Ltd, Wuxi, China) is a new-generation of transient elastography based on a two-dimensional image-guided system to ensure the precise orientation. In the present study, the investigators aim to conduct an international prospective diagnostic trial with 16 sites (Beijing Tsinghua Changgung Hospital, Lanzhou University, The Fifth Medical Center of Chinese PLA General Hospital, Xijing Hospital of Digestive Diseases Wuhan Union Hospital, Zhujiang Hospital, Second Affiliated Hospital of Xi'an Jiaotong University, The Central Hospital of Lishui City, Xingtai People's Hospital, The Seventh Medical Center of Chinese PLA General Hospital Shandong Provincial Hospital, Shunde Hospital, Southern Medical University Medistra Hospital; University of Indonesia, Ankara University School of Medicine, Osaka City University, Chulalongkorn University) to develop and validate the diagnostic performance of FibroTouch-based models for assessing risk of gastroesophageal varices bleeding in compensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years;
* confirmed liver cirrhosis based on liver biopsy or clinical findings;
* compensated liver cirrhosis;
* scheduled to undergo esophagogastroduodenoscopy;
* estimated survival time> 24 months, and model for end-stage liver disease (MELD) score< 19;
* with written informed consent.

Exclusion Criteria:

* contradictions for esophagogastroduodenoscopy;
* body mass index> 35 kg/m2;
* presence of decompensation events (e.g. ascites, variceal bleeding, hepatic encephalopathy, etc.);
* previous esophageal variceal banding legation or transjugular intrahepatic portosystemic shunt;
* current use of non-selective beta-blockers;
* with portal vein thrombosis or hepatocellular carcinoma;
* non-cirrhotic portal hypertension;
* pregnancy or unknown pregnancy status.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with compensated liver cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-12-14 (Actual); Primary Completion 2021-06-13 (Actual); Study Completion 2022-03-13 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of FibroTouch-based models for the risk of variceal bleeding | 1 day
  Diagnostic accuracy of FibroTouch-based models to determine the high-risk or low-risk of variceal bleeding with esophagogastroduodenoscopy as the reference standard

SECONDARY OUTCOMES:
The correlation between FibroTouch-based models and HVPG | 1 day
  The correlation between FibroTouch-based models and hepatic venous pressure gradient (HVPG)
Diagnostic accuracy of FibroTouch-based models for the decompensated events of cirrhotic portal hypertension | 1 year
  Diagnostic accuracy of FibroTouch-based models to determine the presence or absence of decompensated events (e.g. first variceal bleeding) within 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jiahong Dong, MD, Principal Investigator — Beijing Tsinghua Changgeng Hospital; Xiaolong Qi, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (16):
- China (12):
  - The Seventh Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The Fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital of Tsinghua University, Beijing, Beijing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Shunde Hospital, Southern Medical University, Shunde, Guangdong
  - Xingtai People's Hospital, Xingtai, Hebei
  - Wuhan Union Hospital, China, Wuhan, Hubei
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xian, Shanxi
  - Xijing Hospital of Digestive Diseases, Xi’an, Shanxi
  - The Central Hospital of Lishui City, Lishui, Zhejiang
- Medistra Hospital, University of Indonesia, Jakarta, Indonesia
- Osaka City University, Osaka, Japan
- Department of Medicine, Chulalongkorn University, Bangkok, Thailand
- Ankara University School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Undecided.

REFERENCES:
- [Background] Qi X, Berzigotti A, Cardenas A, Sarin SK. Emerging non-invasive approaches for diagnosis and monitoring of portal hypertension. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):708-719. doi: 10.1016/S2468-1253(18)30232-2. PMID 30215362
- [Background] Liu F, Ning Z, Liu Y, Liu D, Tian J, Luo H, An W, Huang Y, Zou J, Liu C, Liu C, Wang L, Liu Z, Qi R, Zuo C, Zhang Q, Wang J, Zhao D, Duan Y, Peng B, Qi X, Zhang Y, Yang Y, Hou J, Dong J, Li Z, Ding H, Zhang Y, Qi X. Development and validation of a radiomics signature for clinically significant portal hypertension in cirrhosis (CHESS1701): a prospective multicenter study. EBioMedicine. 2018 Oct;36:151-158. doi: 10.1016/j.ebiom.2018.09.023. Epub 2018 Sep 27. PMID 30268833
- [Background] Wang FS, Fan JG, Zhang Z, Gao B, Wang HY. The global burden of liver disease: the major impact of China. Hepatology. 2014 Dec;60(6):2099-108. doi: 10.1002/hep.27406. Epub 2014 Oct 29. PMID 25164003
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Berzigotti A, Seijo S, Arena U, Abraldes JG, Vizzutti F, Garcia-Pagan JC, Pinzani M, Bosch J. Elastography, spleen size, and platelet count identify portal hypertension in patients with compensated cirrhosis. Gastroenterology. 2013 Jan;144(1):102-111.e1. doi: 10.1053/j.gastro.2012.10.001. Epub 2012 Oct 8. PMID 23058320
- [Background] Bhardwaj A, Kedarisetty CK, Vashishtha C, Bhadoria AS, Jindal A, Kumar G, Choudhary A, Shasthry SM, Maiwall R, Kumar M, Bhatia V, Sarin SK. Carvedilol delays the progression of small oesophageal varices in patients with cirrhosis: a randomised placebo-controlled trial. Gut. 2017 Oct;66(10):1838-1843. doi: 10.1136/gutjnl-2016-311735. Epub 2016 Jun 13. PMID 27298379
- [Background] Zhu Q, Wang W, Zhao J, Al-Asbahi AAM, Huang Y, Du F, Zhou J, Song Y, Xu K, Ye J, Yang L. Transient Elastography Identifies the Risk of Esophageal Varices and Bleeding in Patients With Hepatitis B Virus-Related Liver Cirrhosis. Ultrasound Q. 2018 Sep;34(3):141-147. doi: 10.1097/RUQ.0000000000000373. PMID 30020268
- [Background] Qi X, An W, Liu F, Qi R, Wang L, Liu Y, Liu C, Xiang Y, Hui J, Liu Z, Qi X, Liu C, Peng B, Ding H, Yang Y, He X, Hou J, Tian J, Li Z. Virtual Hepatic Venous Pressure Gradient with CT Angiography (CHESS 1601): A Prospective Multicenter Study for the Noninvasive Diagnosis of Portal Hypertension. Radiology. 2019 Feb;290(2):370-377. doi: 10.1148/radiol.2018180425. Epub 2018 Nov 20. PMID 30457484